CLINICAL TRIAL: NCT07083713
Title: Group Coaching for Life Goals in People With Neurological Conditions: A Feasibility Study
Brief Title: Group Coaching Study for Life Goals
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRIS-ID-2024-1010
Record Dates: First submitted 2025-06-26; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Students; Spinal Cord Injury; Ehlers Danlos Syndrome; Care Givers
MeSH Terms: conditions — Spinal Cord Injuries; Ehlers-Danlos Syndrome

STUDY DESIGN:
Intervention Model Description: Feasibility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group coaching (Experimental): Group coaching 10 sessions
  Interventions: Behavioral: Group Coaching

INTERVENTIONS:
Behavioral: Group Coaching — Group coaching using a protocol developed with Coaching in Context model

SUMMARY:
This study plans to implement's group coaching with neurodivergent STEM undergraduate students, individuals with spinal cord injuries and their caregivers, and individuals with Ehler's Danlos Syndrome. A trained coach will facilitate the 10 group coaching sessions using the project created coaching protocol. Assessments at pretest and posttest will include two measures addressing the concept of self-efficacy and two others addressing belonging, as well as a battery of tools estimating feasibility.

DETAILED DESCRIPTION:
Background Individuals who have chronic conditions which impact their participation in daily activities generally experience reduced self-efficacy and belonging, which are known to affect their quality of life. Building capacity in these areas is possible as evidenced by the group peer mentoring literature, the individual coaching literature, and the outcomes of Jefferson's GOALS2 program. Group coaching combines the key features of these two approaches but has yet to be used to build capacity in these groups.

Objective To examine group coaching's feasibility and utility for building self-efficacy and belonging.

Hypothesis Group Coaching will increase self-efficacy and belonging by a change effect of 20% as per the General Self-Efficacy Scale, Relationship Closeness Scale, and the Sense of Belonging Scale.

Inclusion criteria People with four types of chronic conditions are included.

1. Neurodivergent students:

   Jefferson neurodivergent undergraduate STEM students Jefferson students who major in Chemistry, Biochemistry, Biology, Pre-Medical Studies, Psychology/biopsychology, Textiles production science, Industrial design, Engineering, Health Sciences, or Exercise science
2. Ehler's Danlos Syndrome:

   * Have been diagnosed by a physician with any form of Ehlers-Danlos Syndromes
   * understand and speak English fluently
   * Be a resident of the United States.
   * be 18 years of age and older
   * has the ability to join the group coaching session by phone or video conferencing.

     3 Person with SCI:
   * Self-report as having a spinal cord injury or disease
   * Understand and speak English fluently
   * Be a resident of the United States.
   * Be 18 years of age and older
   * Stable health condition
   * Have the ability to join the group coaching session by phone or video conferencing. 4 Care partner of a Person with SCI:
   * Provides part or full-time care for a family member/significant other with SCI, need not live in the same household Understand and speak English fluently
   * Be a resident of the United States.
   * Be 18 years of age and older
   * Stable health condition
   * Have the ability to join the group coaching session by phone or video conferencing.

Procedures Recruitment will involve flyers online on websites, social media, newsletters, patient portals, support groups, clinics, and hospitals. Research staff will then reach out to the participant to schedule the COPM over zoom. The zoom meeting will start with the OHR-8H form to confirm the participants willingness to participate. After consenting, the participant will provide information for the COPM, which will be recorded by the research staff member. After completion of the COPM, the participant is provided with a Jefferson Qualtrics link to the following surveys: Social demographic questionnaire General Self-Efficacy Scale, Relationship Closeness Scale, and the Sense of Belonging Scale. The surveys are completed during the zoom call with the research staff member present to answer any questions the participant may have while completing the surveys. After survey completion, participants will be asked to provide their avalability for the group coaching session. After research staff have selected a date for the coaching session, participants will be sent an email informing them of the time and the topic of the coaching session. A reminder email will be sent 24 hours before the session. A total of 10 group coaching sessions will occur for each participant. These will occur in two groups of up to six participants each. The coaching sessions will include conversations regarding specific topics with the goal of facilitating participant in gaining insight and strategies towards set goal. The goals are based on the earlier COPM interview. The coaching sessions will be facilitated by two trained coaches who are study staff members. These coaching sessions will be audio recorded over zoom. Research staff will later fill out surveys including the AIM, IAM, & FIM based on their experiences will the coaching sessions. After the completion of the 10 coaching sessions, participants are scheduled for a second COPM over zoom. The participant will assess their progress based on their earlier COPM, and the interview will be recorded by the research staff member. After completion of the COPM, the participant is provided with a Jefferson Qualtrics link to the following surveys: General Self-Efficacy Scale, Relationship Closeness Scale, the Sense of Belonging Scale, and to determine feasibility through the Acceptability of Intervention Measure (AIM), Feasibility of Intervention Measure (FIM), and Intervention Appropriateness Measure (IAM). The surveys are completed during the zoom call with the research staff member present to answer any questions the participant may have while completing the surveys. After survey completion, the participant will be thanked for their time and a time will be scheduled for picking up their ClinCard payment.

Analysis Demographic data will be summarized descriptively, mean, and standard deviation scores for the intervention feasibility and percentage of completion for the assessment will be determined for assessment of feasibility. Assessment of the outcome measures will be done to calculate how many participants reached the change effect of 20%. Satisfaction will also be assessed using descriptive statistics. Qualitative analysis will be conducted on the session transcripts. Feasibility will be assessed using the AIM, IAM, & FIM.

ELIGIBILITY:
Inclusion Criteria:

* People with four types of chronic conditions are included.

  1. Neurodivergent students:

     Jefferson neurodivergent undergraduate STEM students Jefferson students who major in Chemistry, Biochemistry, Biology, Pre-Medical Studies, Psychology/biopsychology, Textiles production science, Industrial design, Engineering, Health Sciences, or Exercise science
  2. Ehler's Danlos Syndrome:

     * Have been diagnosed by a physician with any form of Ehlers-Danlos Syndromes
     * understand and speak English fluently
     * Be a resident of the United States.
     * be 18 years of age and older
     * has the ability to join the group coaching session by phone or video conferencing.

       3 Person with SCI:
     * Self-report as having a spinal cord injury or disease
     * Understand and speak English fluently
     * Be a resident of the United States.
     * Be 18 years of age and older
     * Stable health condition
     * Have the ability to join the group coaching session by phone or video conferencing. 4 Care partner of a Person with SCI:
     * Provides part or full-time care for a family member/significant other with SCI, need not live in the same household Understand and speak English fluently
     * Be a resident of the United States.
     * Be 18 years of age and older
     * Stable health condition
     * Have the ability to join the group coaching session by phone or video conferencing.

Exclusion Criteria:

* Less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | Week 1 and 10
  Performance and Satisfaction is scored for 9 items using a 1 to 10 scoring system, and higher scores indicate better performance and satisfaction.
Acceptability measure | Week 10
  Acceptability of Intervention Measure is scored from 1 to 5, higher scores are better
Feasibility of Intervention measure | Week 10
  Feasibility of intervention is scored from 1 to 5, higher scores are better
Intervention Appropriateness Measure | Week 10
  The appropriateness of the intervention is assessed using this measure. The scoring is from 1 to 5, higher scores are better.

SECONDARY OUTCOMES:
General Self Efficacy | Week 1 and 10
  A measure of self-efficacy has 10 items. The total score is calculated by finding the sum of the all items. The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Relationship Closeness Scale | Week 1 and 10
  Peers in group and with others are measured on this scale from 1 to 7, and higher scores are better.
Sense of Belonging | Week 1 and 10
  A measure that assesses the sense of belonging in a group, higher scores are better. Each item is scored from 1 to 4, mean scores calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Cadematori C, Alpajora B, Sivori T, Betz S, Gerhardt N, Dunn W, Mulcahey MJ. Preliminary examination of Coaching in Context with clients with spinal cord injury. Spinal Cord Ser Cases. 2021 Apr 13;7(1):27. doi: 10.1038/s41394-021-00391-9. PMID 33850100
- [Background] Mulcahey MJ, Gerhardt N, Alpajora B, Thielen CC, Dunn W. Coaching-in-Context With Informal Maternal Care Partners of Children With Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2022 Winter;28(1):99-113. doi: 10.46292/sci21-00045. Epub 2022 Jan 19. PMID 35145338
- [Background] Potvin MC, West EK, Morales AN, Sailor KS, Coronado N. "I Could Really Use This": Occupational Therapy Students' Perceptions of Learning to Coach. Occup Ther Int. 2022 Oct 13;2022:2266326. doi: 10.1155/2022/2266326. eCollection 2022. PMID 36312841